CLINICAL TRIAL: NCT02210286
Title: The Use of Magnesium L-Threonate for the Enhancement of Learning and Memory in People With Mild to Moderate Dementia
Brief Title: Magnesium L-Threonate for the Enhancement of Learning and Memory in People With Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Magceutics, Inc. (Industry)
Responsible Party: Principal Investigator, Natalie Rasgon, Professor, Director of Center for Neuroscience in Women's Health, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 29329
Record Dates: First submitted 2014-08-01; First posted 2014-08-06 (Estimated); Results first posted 2021-02-02 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Dementia; Alzheimer's Disease
Keywords: dementia; magnesium; learning; memory; Alzheimer's disease
MeSH Terms: conditions — Dementia; Alzheimer Disease | interventions — threonic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Magtein (Experimental): All participants will orally take a total of 1800 mg/day for 60 days. Oral administration includes two pills 2 hours before bed time and one pill in the morning, each pill containing 600 mg of MgT-1219.
  Interventions: Dietary Supplement: Magtein

INTERVENTIONS:
Dietary Supplement: Magtein
  Other Names: magnesium l-threonate

SUMMARY:
The purpose of this study is to examine the effects of supplementing Magnesium L-Threonate in people with mild to moderate dementia. The investigators' goal is to understand whether Magnesium L-Threonate will be associated with improvement in memory and brain function.

DETAILED DESCRIPTION:
Emerging research on the effects of a novel magnesium compound of L-Threonic Acid Magnesium Salt (L-TAMS) containing Vitamins C and D on cognitive performance suggests that supplementation may benefit individuals with Alzheimer's disease (AD). This proof of concept will assess whether supplementation with Magtein (MGT), a constant release formula of Magnesium L-threonate, Vitamin C, and Vitamin D, is associated with changes in regional cerebral metabolism in elderly people with mild to moderate dementia.

This is an open-label, two-month trial consisting of 15-20 participants aged 60 and older with mild to moderate dementia. Subjects will receive 1,800 mg/day of MgT-1219 for a total of 60 days. They will be given neurocognitive testing, blood chemistries, and FDG-PET imaging at baseline, 60 days and more testing at 180 days to assess the acute effect of MgT-1219 on hippocampal and PFC-mediated executive function, attention, reasoning, and memory. Blood draws will be conducted prior to treatment initiation to assess kidney and liver function, complete blood count, fasting plasma insulin, and red blood cell magnesium.

Our outcome measures include a combination of neuropsychological testing and neuroimaging. These will be employed to measure changes in the degree of cognitive impairment within subjects over time, as well as between subjects in the intervention and control groups. FDG-PET imaging will be used to assess the degree of synaptic activity and density within subjects at different time points in the study. These measures will be supplemented by measures of, sleep quality, daytime sleepiness, depression, and activities of daily living.

ELIGIBILITY:
Inclusion Criteria:

* People of either gender > 60 years of age.
* Subject scores between 16 and 26 on the MMSE
* Subject or representative is willing to sign the consent for prior to enrollment into the study and to participate in all aspects of the study. Prospective subject must give verbal assent if unable to sign written consent.
* Adequate visual and auditory acuity to allow neuropsychological testing.
* Greater than 12 years of educational achievement, or a General Education Development certificate to allow adequate neuropsychological testing, and consistency of sample.
* Female subject is surgically sterile, post-menopausal or agrees to use an acceptable method of birth control.
* Subject agrees to stop taking any vitamins, minerals, or dietary/herbal supplements he/she is currently taking at least 7 days prior to randomization and agrees to not take any vitamins, minerals or dietary/herbal supplements other than the study product until after study completion.

Exclusion Criteria:

* Active heart disease
* Uncontrolled high blood pressure (≥ 140/90 mmHg)
* Renal or hepatic impairment/disease
* Type I diabetes
* Unstable thyroid disease
* Psychiatric disorder (hospitalized in the past year)
* History of drug or alcohol abuse.
* Immune disorder (such as HIV/AIDS)
* TIAs, carotid bruits, or verified lacunes
* Significant pulmonary disease
* Contraindication for a PET scan including those who have had a stroke or heart attack in the past 6 months, and those unable or unwilling to lie down for 1 hour.
* Any medical condition deemed exclusionary by the Principal Investigator (PI)
* History of cancer (except localized skin cancer without metastases or in situ cervical cancer) within 5 years prior to screening.
* Currently taking any medications that are known to interact with magnesium.
* Currently taking antibiotics as the study product may reduce the absorption of antibiotics. A washout period of 2 weeks is allowed.
* On an unstable dose of medication (defined as fewer than 90 days at the same dose).
* Currently taking any medication deemed exclusionary by PI.
* Allergy or sensitivity to any ingredient in the test product.
* Evidence of hepatic or renal dysfunction
* History of drug or alcohol abuse in the past 12 months.
* Pregnant , lactating, or planning to become pregnant during the study period.
* Subject has any condition or abnormality that, in the opinion of the investigator, would compromise the safety of the subject or the quality of the study data.
* Subject is participating or has participated in another research study within 30 days prior to the screening visit.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2014-07; Primary Completion 2016-04 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Natalie L Rasgon, MD, Ph.D, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Department of Psychiatry & Behavioral Sciences, Stanford, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Magtein: 17 subjects were then enrolled into the study
Period: Overall Study
Arm/Group | Magtein
Started | 17
Completed | 15
Not Completed | 2

BASELINE CHARACTERISTICS:
Groups:
- Magtein Subjects: Inclusion criteria included adults of either gender > 60 years of age (women had to be post-menopausal), a diagnosis of probable AD from their physician, a Mini-Mental State Examination (MMSE) between 14 and 24, adequate visual and auditory acuity to allow for neuropsychological testing, at least 12 years of education (or a GED to allow consistency of the sample), and willingness to or having a representative willing to sign the informed consent prior to enrollment into the study (for those subjects unable to sign or understand informed consent, assent to participate in the study was required), and agreeing to discontinue vitamins, minerals, or dietary/herbal supplements for at least 7 days prior to study entry and until after study completion.
Arm/Group | Magtein Subjects
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 77.0 (5.86)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Two participants discontinued the intervention before analysis
  Participants
    number analyzed (Participants) | 15
    Female | 7
    Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Cognitive Function
Description: Neurocognitive assessment - Domain-specific composite scores for the four following cognitive areas include:
  1a) Alzheimer's Disease Assessment Scale - cognitive subscale (ADAS-COG) (min: 0, max: 70, higher = better, units on a scale)
  1b) Mini Mental Status Examination (MMSE) (min: 0, max : 30, higher = better, units on a scale)
  1c) Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) (min: 40, max: 160, higher = better, units on a scale)
  1d) Wechsler Adult Intelligence Scale - Fourth edition (WAIS-IV) (min: 85 , max: 115, higher = better, units on a scale)
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Magtein Cognitive Data: Participants were assessed with the ADAS-Cog, MMSE, D-KEFS RBANS, and WAIS-IV neuropsychological assessments. We hypothesized improvements in cognitive scores with MMFS-201-101 treatment.
Arm/Group | Magtein Cognitive Data
Number analyzed (Participants) | 17
units on a scale
  ADAS-COG | -0.58 (7.58)
  MMSE | -1.73 (2.49)
  RBANS | -0.36 (8.83)
  WAIS | -0.07 (1.86)

2. Primary Outcome: Change From Baseline in Cognitive Function (DKEFS Color-Word Test)
Description: 1) Delis-Kaplan Executive Function System Color-Word Test (DKEFS, assesses executive functioning): no minimum or maximum set, higher is worse, total number of errors
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: total number of errors
Groups:
- Change From Baseline in Cognitive Function (DKEFS): Participants were assessed with the ADAS-Cog, MMSE, D-KEFS RBANS, and WAIS-IV neuropsychological assessments. We hypothesized improvements in cognitive scores with MMFS-201-101 treatment.
Arm/Group | Change From Baseline in Cognitive Function (DKEFS)
Number analyzed (Participants) | 17
total number of errors | 0.8 (4.23)

3. Primary Outcome: Change From Baseline in Cognitive Function (DKEFS - Trail 4)
Description: This is a graphomotor test comprised of 5 conditions. Condition 4 (Number Letter Switching) is a measure of cognitive flexibility
Time Frame: Baseline to 6 months
Measure: Mean (Standard Deviation); unit: time in seconds
Groups:
- Change From Baseline in Cognitive Function (DKEFS - Trail 4): Participants were assessed with the ADAS-Cog, MMSE, D-KEFS RBANS, and WAIS-IV neuropsychological assessments. We hypothesized improvements in cognitive scores with MMFS-201-101 treatment.
Arm/Group | Change From Baseline in Cognitive Function (DKEFS - Trail 4)
Number analyzed (Participants) | 17
time in seconds | 23.5 (88.5)

4. Secondary Outcome: Change From Baseline in CMRgl
Description: Brain imaging focusing on the following anatomical regions: medial temporal region (including hippocampus and entorhinal cortex), prefrontal cortex, parietotemporal cortex, posterior cingulate cortex. Increases in the summary index sROI have been shown to track AD-related CMRgl declines.
  We will be focusing on changes in the cerebral metabolic rate for glucose (CMRgl) from baseline to day 67.
Time Frame: Baseline to Day 67
Measure: Mean (Standard Deviation); unit: mmol·min-1·100 g-1
Groups:
- Change in CMRgl From Baseline: We examined CMRgl changes using our summary index statistical region of interest (sROI) which is free of the multiple comparison concern.
Arm/Group | Change in CMRgl From Baseline
Number analyzed (Participants) | 17
mmol·min-1·100 g-1 | 0.0093 (0.031)

5. Secondary Outcome: RBC Magnesium Chemistry
Description: Magnesium (mg/dl) in red blood cells
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: mg/dl
Groups:
- Change in RBC Magnesium: Change in the amount of magnesium in red blood cells (mg/dl) from baseline
Arm/Group | Change in RBC Magnesium
Number analyzed (Participants) | 17
mg/dl | -0.007 (1.16)

ADVERSE EVENTS:
Groups:
- Magtein Adverse Events: See Table below for details on adverse event.
Arm/Group | Magtein Adverse Events
All-Cause Mortality (participants affected / at risk) | 0/17
Serious Adverse Events (participants affected / at risk) | 1/17
Other Adverse Events (participants affected / at risk) | 0/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Magtein Adverse Events (N=17)
GI Problem (Gastrointestinal disorders) | 1 (1) — 1 subject developed mild gastrointestinal discomfort after taking MMFS-201-101

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No